CLINICAL TRIAL: NCT02114632
Title: A Double Blind, Placebo Controlled Trial of Effectiveness of Omega-3 and Omega-6 Polyunsaturated Fatty Acids in Treatment of Children With Attention Deficit/Hyperactivity Disorder
Brief Title: Supplementation of Polyunsaturated Fatty Acids in Children With Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Magdalena Grygo, MD, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: KB/154/2006
Record Dates: First submitted 2014-03-23; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: ADHD
Keywords: ADHD, attention deficit/hyperactivity disorder, attention deficit disorder, inattention, cognitive skills, children, polyunsaturated fatty acids, PUFA
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyunsaturated fatty acids (Active Comparator): 6 capsules of food supplement "Eye q" per day divided in two daily doses (558 mg EPA, 174 mg DHA, 60 mg GLA per day)
  Interventions: Dietary Supplement: Eye Q
- placebo (Placebo Comparator): 6 capsules of olive oil per day divided in two daily doses.

INTERVENTIONS:
Dietary Supplement: Eye Q — 3 months of treatment with a polyunsaturated fatty acids or placebo. At 3 months a one-way treatment crossover of the placebo-group to active treatment was made so that both patient groups received active treatment for the remaining 3 month period.
  Arms: Polyunsaturated fatty acids

SUMMARY:
The purpose of the study is assessing the efficacy of Omega - 3 and Omega - 6 treatment in boys with Attention-Deficit/Hyperactivity Disorder (ADHD) compared with control group healthy boys.

DETAILED DESCRIPTION:
The study is designed as a randomized, double-blind placebo-controlled trial with a total duration of 6 months. 100-120 boys with ADHD aged 8-16 years and 30 healthy boys will will be randomized to 3 months of treatment with a fixed dose of 6 capsules of food supplement "Eye q" per day divided in two daily doses (558 mg eicosapentaenoic acid (EPA), 174 mg docosahexaenoic acid (DHA), 60 mg gamma-linolenic acid (GLA) per day) or to placebo (olive oil). At 3 months a one-way treatment crossover of the placebo-group to active treatment will be made so that both patient groups will receive active treatment for the remaining 3 month period. Control group will receive active treatment for 6 month. The assessment of children will be made 3 times: at the point of start, after 3 months, and after 6 months. The assessments will be made using standardized interviews and questionnaires, neuropsychological tests, pediatric and neurological examination and taking a 5 ml sample of blood to assess level of polyunsaturated fatty acids (PUFA) in serum and in cell membranes of erythrocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be boys between the ages of 8-16 years.
2. Patients must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criteria for ADHD confirmed by Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version (K-SADS-PL)
3. Patients must be of normal intelligence as assessed by the Wechsler Intelligence Scale for Children - Revised Edition (WISC-R).
4. Treatment of ADHD by such drugs as: atomoxetine, reboxetine, clonidine, desipramine or clomipramine or children with ADHD without pharmacological treatment

Exclusion Criteria:

1. Patients who have a documented history of Bipolar I or II disorder, psychosis or autism.
2. Patients with a history of epilepsy
3. Patients with a history of asthma treated with corticosteroids.
4. Patients with diabetes, haemorrhagic problem, hyperlipidemia, hypertension, hyperthyroidism or hypothyroidism.
5. Patients taking any psychotropic medication other than above-mentioned on a regular basis, including health-food supplements that the investigator feels have central nervous system activity, must have a washout equal of at least three months before study entry, and such medications are not allowed during the study.
6. Patients with a history of alcohol or drug abuse within the past 3 months (excessive or compulsive use as judged by the investigator).

Ages: 8 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2007-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
assessment of intensity of ADHD symptoms using neuropsychological tests and parents and teacher questionnaires in treated group according to placebo intervention | change from baseline at 6 months

SECONDARY OUTCOMES:
assessment of adverse events. | change from baseline at 6 months

OTHER OUTCOMES:
assessment of connection between level of fatty acids in serum and intensity of ADHD symptoms in treated group according to placebo intervention | change from baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Grygo, MD, Principal Investigator — Medical University of Warsaw, Child and Adolescent Psychiatry Department
Locations (1):
- Child and Adolescent Psychiatry Department, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600